CLINICAL TRIAL: NCT01241162
Title: A Phase I Trial Combining Decitabine and Vaccine Therapy for Patients With Relapsed Neuroblastoma and Sarcoma.
Brief Title: Decitabine Followed by a Cancer Antigen Vaccine for Patients With Neuroblastoma and Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Solving Kids' Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34183
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Neuroblastoma; Ewings Sarcoma; Osteogenic Sarcoma; Rhabdomyosarcoma; Synovial Sarcoma
Keywords: Neuroblastoma; Ewings sarcoma; osteogenic sarcoma; rhabdomyosarcoma; synovial sarcoma; high-risk; relapsed; children
MeSH Terms: conditions — Neuroblastoma; Sarcoma, Ewing; Osteosarcoma; Rhabdomyosarcoma; Sarcoma, Synovial; Recurrence | interventions — Adjuvants, Pharmaceutic; Decitabine; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Experimental): Biological/Vaccine: Autologous dendritic cell vaccine with adjuvant
  Interventions: Biological: Autologous dendritic cell vaccine with adjuvant

INTERVENTIONS:
Biological: Autologous dendritic cell vaccine with adjuvant — Week 1:
  Decitabine (DAC): 10 mg/m2/day IV (Mon-Fri)
  Weeks 2 and 3:
  Vaccine: 3-5 E6 peptide pulsed DC (Mon)
  Hiltonol applied topically to vaccine site before and after vaccination
  Other Names: Decitabine (trade name Dacogen or 5-aza-2'-deoxycytidine/DAC; Hiltonol

SUMMARY:
This treatment study for relapsed high-risk neuroblastoma, Ewings sarcoma, osteogenic sarcoma, rhabdomyosarcoma or synovial sarcoma involves an autologous cancer testis (CT) antigen specific dendritic cell (DC) vaccine preceded by decitabine as a demethylating chemotherapy.

DETAILED DESCRIPTION:
For vaccine production, mature DC will be pulsed with overlapping peptides mixes derived from full-length NY-ESO-1, MAGE-A1, and MAGE-A3.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of relapsed high-risk neuroblastoma,Ewings sarcoma, osteogenic sarcoma, rhabdomyosarcoma, synovial sarcoma
* Patient may have gross tumor that has been treated with multi-agent chemotherapy prior study entry, but does not need to have gross tumor prior to study entry.
* Patients must have had a diagnosis of neuroblastoma or sarcoma either by histological verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
* Have received standard chemotherapy and/or SCT, and are at least 6 months post-transplant.
* Age: Patients must be 1 - < 25 years of age when registered on study.
* Organ Function Requirements: All patients must have adequate organ function defined as:
* Hematological Function: ANC ≥ 500; Platelet count ≥ 75.
* Renal Function: Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 OR A maximum serum creatinine (mg/dL) based on age/gender as follows: 1YO M&F = 0.6, 2-5YO M&F = 0.8, 6-9YO M&F = 1, 10-12YO M&F = 1.2, 13-15YO M = 1.5, 13-15YO F = 1.4, 16+ M = 1.7, 16+ F = 1.4
* Cardiac Function: Patient must have normal cardiac function documented by Ejection fraction (> 55%) documented by echocardiogram or radionuclide MUGA evaluation OR Fractional shortening (≥ 28%) documented by echocardiogram
* Liver Function: Total bilirubin ≤ 1.5 x normal for age, AND SGPT (ALT) and SGOT (AST) ≤ 3 x normal for age.
* Room air pulse oximetry >94%.
* Male and female sexually active patients of reproductive age who wish to participate must agree to use acceptable contraception.
* Lansky performance scale > 70, ECOG < 2 (Appendix I).

Exclusion Criteria:

* Patient is pregnant.
* Patients with a positive result for any of the following diagnostic tests: Hep B Ag, Hep B Core Ab, Hep C Ab, HIV-1 Ab, HIV-2 Ab, HTLV-1 Ab, HTLV-2 Ab, RPR.
* Patient has a history of autoimmune disease, specifically inflammatory bowel disease, systemic lupus erythematosis, or rheumatoid arthritis.
* Patient is receiving concurrent systemic steroid therapy.
* Patient has a known systemic hypersensitivity to DAC, Hiltonol, or any vaccine component.

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2010-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Tolerance of study treatment | 2 years
  Tolerance to DAC, at at least 50% dosing, and 3 of the 4 planned vaccinations during the first two cycles.

SECONDARY OUTCOMES:
Tumor Response | 2 years
  Assessment of tumor responses--complete or partial remission, stable disease, and disease progression--by CT/PET/MIBG or MRI after cycles 2 and 4.
Immune Response | 2 years
  Assessment of post-vaccination T cell responses to MAGE-A1, MAGE-A3, and NY-ESO-1 by immunoassays.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Lucas, MD, Principal Investigator — University of Louisville, Kosairs Charities Pediatric Clinical Research Unit
Locations (1):
- University of Louisville, Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky, United States